CLINICAL TRIAL: NCT03699098
Title: The Incidence and Risk Factors of Radiotherapy Induced Hypothyroidism in Head and Neck Cancer
Brief Title: The Incidence and Risk Factors of Radiotherapy Induced Hypothyroidism in Head and Neck Cancer With Long Term Follow up
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ehab Saad, Principal investigator, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: H&N82017
Record Dates: First submitted 2018-10-02; First posted 2018-10-09 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Head and Neck Cancer
Keywords: hypothyroidism; radiotherapy; head and neck cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Hypothyroidism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: TSH, T3, T4 and thyroid gland DVH — measuring thyroid functions and DVH parameters of thyroid gland

SUMMARY:
This is a retrospective study with long term follow up to evaluate the incidence, timing and risk factors of radiotherapy induced hypothyroidism in non-thyroid head and neck cancer patients who were treated with RT alone or in combination with surgery and/or chemotherapy.

DETAILED DESCRIPTION:
For any patient, fixation was done by a thermoplastic mask. CT scan was done at 3mm thickness for the head and neck region. CT images were transferred to the planning system. Three-dimensional conformal RT, intensity-modulated radiotherapy (IMRT) or Volumetric modulated arc therapy (VMAT) was created. All patients were irradiated with once-daily fractionation at 1.8-2.0 Gy/d with 6-MV photon beams for five days a week. The gross target volume (GTV) was treated with a dose of 70Gy and the lymphatic site (CTV) and areas of high risk microscopic disease (CTV) including lymph nose levels received a radiation dose ranging from 54-66 Gy according to its risk. PTV is a circumferential margin of 5mm around CTV.

Thyroid function parameters:

The patient's serum T4, T3 and TSH levels, were measured during follow up. Clinical hypothyroidism is defined as the increase in TSH above 5.0mIu/ml with a decrease in free thyroxine levels (free T4) in the serum while elevated TSH with normal free T4 levels was labeled as subclinical hypothyroidism .As per institutional values, the normal values intervals of T4 level (7- 25 PMOL/L), T3( 1.5-7 PMOL/L),TSH (0.2-5 mIu/L).

The median time to onset of hypothyroidism was defined as the time interval between completion of radiotherapy and first abnormal recorded T3/T4/TSH value.

For all treated patients, thyroid gland was delineated and by reviewing the DVH, the V45, V50, V55, V60, V65 and V70 which means the volume of the thyroid gland receiving 45 Gy, 50 Gy, 55Gy, 60 Gy and 70 Gy respectively.

ELIGIBILITY:
Inclusion Criteria:

* Non-thyroid head and neck cancer patients who were treated with RT alone or in combination with surgery and/or chemotherapy

Exclusion Criteria:

* Patients with thyroid gland disease or abnormal thyroid hormone levels before radiotherapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-05 (Actual)

PRIMARY OUTCOMES:
The the incidence of hypothyroidism | 8 months
  Measuring the thyroid function tests

SECONDARY OUTCOMES:
The risk factors of hypothyroidism | 8 months
  Defining the risk factors of hypothyroidism

CONTACTS AND LOCATIONS:
Locations (1):
- Department of clinical oncology and nuclear medicine, Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided